CLINICAL TRIAL: NCT03710135
Title: Child Development Resources Investing in Fatherhood: New Pathways - Process Study & Evaluation
Brief Title: CDR Investing in Fatherhood Process Study & Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Child Development Resources (Other)
Responsible Party: Principal Investigator, Laura Parker, Local Evaluator, Child Development Resources
Other Study IDs: 2016/04/2
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Parenting; Parent-Child Relations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the Investing in Fatherhood: New Pathways program of Child Development Resources (CDR), a Healthy Marriage and Responsible Fatherhood (HMRF) grantee. The program will deliver parenting education, relationship skills training, job preparedness and financial planning, and case management support. This research will consist of a descriptive process and program evaluation study, with research questions focusing on recruitment and retention and short-term participant outcomes.

DETAILED DESCRIPTION:
This study will address three research questions:

1. Which recruitment strategies are the most successful for participation? CDR will work to expand recruitment efforts and encourage greater participation through a number of strategies, such as offering various incentives and hosting classes in other spaces (e.g. churches, restaurants, clinics). This study will examine which methods are the most effective.
2. Which engagement/retention strategies are the most successful? Current fatherhood services staff at CDR have expressed difficulty in getting fathers to participate on a regular and steady basis in fatherhood services. CDR will explore several strategies for increased retention and this study will evaluate these strategies.
3. Do fathers who participate in the program earlier in their fatherhood experience (e.g. when their oldest child is under five years of age) report better outcomes than fathers who begin receiving fatherhood services later? CDR has extensive knowledge working specifically with young children and families in early intervention programs. In early childhood development, many studies have shown that the highest return on investment comes from early intervention, from birth through age five. The hypothesis is that this principle holds true in responsible fatherhood programming as well.

ELIGIBILITY:
Inclusion Criteria:

* Any person enrolled in CDR's Pathways Fatherhood program.

Exclusion Criteria:

* Any participant who does not give informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents (majority fathers) who participate in CDR's Pathways Fatherhood program, in the community and incarcerated individuals.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in attitudes toward child | depending on program length, ranges from 30 days to 10 weeks
  nFORM (Information, Family Outcomes, Reporting, and Management) questions on pre- and post-survey. Answers range from (1) Never to (4) Often. A higher response indicates a better outcome.
Change in using negative punishment with child | depending on program length, ranges from 30 days to 10 weeks
  nFORM (Information, Family Outcomes, Reporting, and Management) questions on pre- and post-survey. Answers range from (1) Never to (4) Every Day or Almost Every Day. A lower response indicates a better outcome.
Change in time spent with child | depending on program length, ranges from 30 days to 10 weeks
  nFORM (Information, Family Outcomes, Reporting, and Management) questions on pre- and post-survey. Answers range from (1) Never to (4) Every Day or Almost Every Day. A higher response indicates a better outcome.
Change in feeling overwhelmed with parenting responsibilities | depending on program length, ranges from 30 days to 10 weeks
  nFORM (Information, Family Outcomes, Reporting, and Management) questions on pre- and post-survey. Answers range from (1) Never to (4) Often. A lower response indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Child Development Resources, Williamsburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No